CLINICAL TRIAL: NCT00607360
Title: Integration of the Therapeutic Workplace in Drug Court
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Conrad J. Wong, Ph.D./ Assistant Professor, University of Kentucky College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-0865-F2L; 7R21DA017885-02 (NIH)
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2008-01

CONDITIONS: Drug Addiction
Keywords: cocaine addiction, treatment, contingency management, employment intervention
MeSH Terms: conditions — Substance-Related Disorders; Cocaine-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Drug Court (No Intervention): Participants received standard services from drug court
- Drug Court plus Therapeutic Workplace (Experimental): Participants receive standard drug court services plus therapeutic workplace intervention
  Interventions: Behavioral: Therapeutic Workplace Intervention

INTERVENTIONS:
Behavioral: Therapeutic Workplace Intervention — Therapeutic workplace intervention is intended for individuals with drug addiction and chronic unemployment. Participants are invited to participate in work and receive salary for participation and productivity contingent upon drug abstinence.
  Arms: Drug Court plus Therapeutic Workplace

SUMMARY:
Drug Courts were developed as a therapeutic alternative to incarceration of drug-involved offenders by providing 'judicially supervised' drug abuse treatment and probation for nonviolent offenders in lieu of criminal prosecution and incarceration. Outcome studies have shown that drug courts have modest effects on participation in drug abuse treatment, drug use, and employment. The Therapeutic Workplace intervention is an effective employment-based treatment that integrates abstinence reinforcement contingencies in a work setting, intended to treat individuals with histories of drug addiction and chronic unemployment. Under this intervention, drug abuse patients are hired and paid to work. To promote abstinence, patients are required to provide drug-free urine samples to gain and maintain daily access in the workplace. In this way, patients can work and earn salary, but only as long as they remain drug abstinent. Patients using drugs and lacking job skills participate in an initial training phase to initiate abstinence and establish computer data entry skills. Once abstinent and skilled, patients are hired into an income-producing Therapeutic Workplace data entry business. Given that many drug court participants suffer from long histories of drug addiction and unemployment, the Therapeutic Workplace could be ideal for this population. This proposes of this clinical trial is to evaluate the Therapeutic Workplace intervention in a Drug Court.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Drug Court
* Report using any opiates and/or cocaine during 30 days prior to their arrest
* Unemployed

Exclusion Criteria:

Individuals are excluded if they:

* Are at imminent risk of suicide
* Have a psychotic disorder that may limit their workplace functioning or their ability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2004-08; Study Completion 2007-07 (Actual)